CLINICAL TRIAL: NCT01362309
Title: D-Cycloserine to Enhance Extinction to Alcohol Cues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Boston University (Other); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R21AA017696 (NIH); R21AA017696 (NIH)
Record Dates: First submitted 2011-05-24; First posted 2011-05-30 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2011-05

CONDITIONS: Alcohol Use Disorders.
Keywords: Alcohol; Cues; Extinction; D-Cycloserine
MeSH Terms: conditions — Alcoholism | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Inert filler in matched pill.
  Interventions: Drug: d-cycloserine.
- d-cycloserine 50 mg (Active Comparator): 50 mg d-cycloserine.
  Interventions: Drug: d-cycloserine.

INTERVENTIONS:
Drug: d-cycloserine. — 50 mg administered on two occasions.
  Other Names: Seromycin.

SUMMARY:
There is considerable evidence that Alcohol Use Disorders (AUDs) can be understood as a form of dysregulated learning and are influenced by classical conditioning. This is based on numerous studies indicating that conditioned contextual cues influence craving for alcohol consumption. As a result, there has been considerable interest in extinction-based treatments for AUDs (i.e., treatments that focus on extinguishing the associations between alcohol cues and motivation to drink), referred to as cue exposure treatment To date, extinction-based treatment for AUDs has resulted in disappointing outcomes in clinical trials and there is considerable interest in improving this form of treatment. One novel strategy is the use of pharmacological adjuncts to enhance extinction. Medications that maximize extinction may minimize subsequent reactions to alcohol cues and, in turn, subsequent clinical outcomes. This study is examining whether the medication d-cycloserine (DCS) can enhance extinction to alcohol cues. Recent basic research has revealed that DCS enhances extinction to fear cues and several lines of evidence suggest that DCS may also enhance extinction to alcohol cues. Therefore, DCS may serve as a useful pharmacological adjunct to extinction-based treatment for AUDs. Our primary aim is to examine whether, compared to placebo, DCS (50 mg) will enhance extinction to alcohol cues under controlled laboratory conditions in treatment-seeking individuals with alcohol use disorders. We hypothesize that DCS will generate greater extinction compared to placebo during the subsequent extinction session as measured by attenuated craving in response to alcohol cues. Furthermore, we hypothesize that DCS will generate greater extinction compared to placebo at follow-up assessments. This study is a proof-of-concept test of whether DCS can reduce reactions to alcohol cues under controlled laboratory conditions. It is a preliminary study using a subclinical number of extinction sessions and medication administrations to establish whether or not DCS improves extinction in the laboratory. If proof-of-concept is supported, it will suggest that a clinical trial is warranted. A clinical sample and clinical context are used to maximize the potential generalizability from this exploratory study.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of an alcohol use disorder.
2. At least 14+/7+ drinks/week for males/females.
3. Alcohol cue reactivity.
4. 9th grade education or greater.
5. 21-65 years old.
6. Stable contact information.
7. Treatment-seeking.

Exclusion Criteria:

1. Participation in a previous study of d-cycloserine.
2. Mandated to treatment.
3. Significant withdrawal symptoms (i.e., Clinical Institute Withdrawal Scale - Revised score of 15+, history of previous withdrawal-related hospitalizations, or withdrawal-related hallucinations).
4. Current DSM IV Axis I conditions other than alcohol and nicotine dependence.
5. Living with a previous study participant.
6. No medical contraindications for d-cycloserine (i.e., currently taking ethionamide, isoniazid, SSRIs, history of epilepsy, history of hypersensitivity to DCS, or additional medical conditions deemed a risk at the physical exam by a study physician).
7. Cardiovascular disease or uncontrolled hypertension (such conditions may contribute to abnormal psychophysiological arousal data), as determined by the study physician.
8. Pregnant or seeking to conceive (females only).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in Craving for alcohol. | Laboratory sessions (two, one-week apart): change in craving over 11 occasions, 5 minutes apart. Between sessions: change in craving across 7 occasions (Study Day: 1, 4, 7, 12, 19, 33, 40).
  Subjective desire for alcohol is assessed intermittently during extended exposure to alcohol cues with response prevention within laboratory sessions and over the preceding week at 6 study visits.

SECONDARY OUTCOMES:
Change in Tolerability | Prevalence and change in side effects measured on 4 occasions (Study Day: 1, 4, 7, 12)
  Side effects resulting from d-cycloserine in individuals with alcohol use disorders.

CONTACTS AND LOCATIONS:
Overall Officials: James MacKillop, PhD, Principal Investigator — University of Georgia
Locations (1):
- Experimental and Clinical Psychopharmacology Laboratory, Dept. of Psychology, University of Georgia, Athens, Georgia, United States